CLINICAL TRIAL: NCT02020317
Title: Clinical Decision Support System for Quality Assurance in Potassium-Increasing Drug-Drug-Interactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FZMI-KEK-ZH-Nr. 2013
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Hyperkalemia
Keywords: drug interactions; Drug Monitoring; Potassium; Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- computer-based reminders and alerts (Active Comparator): Behavioral: display of computer-based reminders for serum potassium monitoring and hyperkalemia alerts (decision support in potassium-inc. drug-drug-interactions)
  Interventions: Behavioral: decision support in potassium-inc. drug-drug-interactions
- no computer-based reminders or alerts (No Intervention): Behavioral: no display of computer-based reminders for serum potassium monitoring and hyperkalemia alerts

INTERVENTIONS:
Behavioral: decision support in potassium-inc. drug-drug-interactions — display of computer-based reminders for serum potassium monitoring and hyperkalemia alerts
  Arms: computer-based reminders and alerts

SUMMARY:
To investigate the impact of reminders for serum potassium monitoring and of hyperkalemia alerts during potassium-increasing drug-drug-interactions.

DETAILED DESCRIPTION:
The development of hyperkalemia during potassium-increasing drug-drug-interactions (DDIs) is associated with (i) unknown or elevated serum potassium level at onset of treatment and (ii) insufficient monitoring of serum potassium during therapy. However, potassium-increasing DDIs are frequently started despite an unknown or elevated serum potassium level, and monitoring intervals often exceed 48 hours.

This study investigates the impact of reminders for serum potassium monitoring and hyperkalemia alerts. Both reminders and alerts are displayed in the electronic patient chart of in-patients treated with potassium-increasing DDIs.

ELIGIBILITY:
Inclusion criteria:

* in-patients treated with concurrent potassium-increasing drugs

Exclusion criteria:

* outpatients; in-patients on wards without computerized physician order entry (i.e. patients treated in the ICU)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3341 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Impact on serum potassium monitoring during potassium-increasing drug-drug-interactions | 1 year
  Rate of serum potassium monitoring intervals of < = 72 hours during potassium-increasing drug-drug-interactions in proportion to all serum potassium monitoring intervals during potassium-increasing drug-drug-interactions

SECONDARY OUTCOMES:
Frequency of hyperkalemia during potassium-increasing drug-drug-interactions | 1 year
Frequency of potassium-increasing drug-drug-interactions ordered in the presence of hyperkalemia | 1 year
Frequency of transfers to the ICU during potassium-increasing drug-drug-interactions in function of the serum potassium level | 1 year
Frequency of death during potassium-increasing drug-drug-interactions in the presence or absence of hyperkalemia | 1 year
Change in frequency distribution of serum potassium monitoring intervals | 1 year
Response of physicians to the computer-based alerts and reminders | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Blaser, PhD, Prof, Principal Investigator — University Hospital Zurich, Center for Clinical Research, Research Center for Medical Informatics
Locations (1):
- University Hospital Zurich, Center for Clinical Research, Research Center for Medical Informatics, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Eschmann E, Beeler PE, Kaplan V, Schneemann M, Zund G, Blaser J. Patient- and physician-related risk factors for hyperkalaemia in potassium-increasing drug-drug interactions. Eur J Clin Pharmacol. 2014 Feb;70(2):215-23. doi: 10.1007/s00228-013-1597-2. Epub 2013 Oct 23. PMID 24150532
- [Background] Eschmann E, Beeler PE, Zund G, Blaser J. Evaluation of alerts for potassium-increasing drug-drug-interactions. Stud Health Technol Inform. 2013;192:1056. PMID 23920830